CLINICAL TRIAL: NCT00206752
Title: A Randomized Prospective Evaluation of Unilateral/Ipsilateral Neck Irradiation in Selected Patients With Squamous Cell Carcinoma of the Head and Neck Who Are Managed by Radiation Therapy
Brief Title: Study of Unilateral Neck Irradiation in Patients With SCC of the Head and Neck
Acronym: Unilateral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 186-03; ETH136-03D
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

ARMS (1):
- unilateral radiation therapy (Experimental): definitive external beam radiation in the ipsilateral neck.
  Interventions: Radiation: Radiation therapy; Radiation: definitive external beam radiation in the ipsilateral neck

INTERVENTIONS:
Radiation: Radiation therapy — definitive external beam radiation in the ipsilateral neck.
Radiation: definitive external beam radiation in the ipsilateral neck — definitive external beam radiation in the ipsilateral neck

SUMMARY:
The purpose of this study is to assess the feasibility of avoiding opposite side neck radiation therapy in patients with clearly one side squamous cell cancer of the head and neck. We aim to assess the reduction in treatment volume (amount of radiation therapy required), and the resultant xerostomia and mucositis, with the delivery of unilateral neck radiation therapy.

DETAILED DESCRIPTION:
Patients will be treated with definitive external beam radiation plus/minus chemotherapy plus/minus neck dissection in the ipsilateral neck (post radiation). The primary site will be treated with definitive radiation therapy, or definitive surgery plus post-operative radiation therapy. Primary endpoints are loco-regional control, as well as quality of life, xerostomia, mucositis, and neck fibrosis.

Salivary evaluations shall be performed prior to the initiation of radiation therapy, during the second week of EBRT, and at the completion of radiation. Evaluations will also be conducted at 3, 6, and 12 months after the completion of EBRT.

Oral mucositis will be assessed prior to the initiation of EBRT and weekly during EBRT. Evaluations will also be conducted at 3 and 6 months after the completion of EBRT. Two standardized mucositis scales will be used: the RTOG scale and the WHO scale.

Clinical response will be evaluated by physical exam and PET/CT. PET/CT scans will be done at 3, 6, 12, 18, and 24 months, and then when clinically indicated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the oral cavity or oropharynx, with the primary lesion >1 cm from the midline.
* Patient has no clinical or radiologic evidence of contralateral neck node metastases.
* No evidence of distant metastasis.
* No previous history of radiation therapy or chemotherapy
* performance status 0-2
* Age >= 18
* Signed informed consent
* Patients must be accessible for treatment and follow-up

Exclusion Criteria:

* HIV positive patients
* Pregnancy or any patients not practicing contraception
* Active tobacco or alcohol addiction (as assessed by medical caregiver)
* Serious comorbid disease which prevents delivery of full treatment including psychiatric disorders, cardiopulmonary disease, etc.
* Concomitant use of any trial anticancer therapeutic within 30 days of entry
* Uncontrolled hypertension
* Known hypersensitivity to mammalian cell-derived products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
FACT (head and neck);Xerostomia related Quality of Life Questionnaire | September 2010

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hu, MD, Principal Investigator — Department of Radiation Oncology at Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States